CLINICAL TRIAL: NCT05757895
Title: Investıgatıon of the Effect of Trunk dısorder Level on partıcıpatıon, actıvıty and qualıty of lıfe Level of chıldren wıth Cerebral Palsy at prımary School Level
Brief Title: Investigation of Trunk Control in Spatic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, PhD, Karabuk University
Other Study IDs: Cerebral Palsy
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy, trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiparetic SP: The Level of Gross Motor Function Classification System (GMFCS), Trunk Affect Level ( Trunk Impairment Scale- TIS), Activity Level ( Gross Motor Function Criterion- GMFM-88), Participation Level ( Pediatric Data Collection Tool- PODCI) and Quality of Life Level (Cerebral Palsy Questionnaire for Children Cerebral Palsy Module- PedsQL) will be evaluated.
- Diparetic SP: The Level of Gross Motor Function Classification System (GMFCS), Trunk Affect Level ( Trunk Impairment Scale- TIS), Activity Level ( Gross Motor Function Criterion- GMFM-88), Participation Level ( Pediatric Data Collection Tool- PODCI) and Quality of Life Level (Cerebral Palsy Questionnaire for Children Cerebral Palsy Module- PedsQL) will be evaluated.

SUMMARY:
Cerebral Palsy is a disease characterized by movement, posture and tone disorders that occur in the immature brain structure that has not yet completed its development anatomically and physically, but can undergo permanent changes. Although the prevalence is 2-3/1000 births, this rate is 4.4/1000 births in our country. As the level of development of the country increases, this rate decreases. Cerebral Palsy is clinically classified according to different criteria and types. While the terms hemiplegia, diplegia, tetraplegia are used according to limb involvement, terms such as spastic, ataxic, dyskinetic, hypotonic are used in classification according to dominant tone disorders.

Postural control, which plays a key role in the realization of all our fine and gross motor skills and is necessary for the realization of our daily life activities, is insufficient in children with cerebral palsy, a neurological disorder. Insufficient postural control negatively affects mobility, limb movements, static and dynamic trunk control.

When the literature is scanned and trunk postural control more of the physical/motor, we investigated the effect of parameters, which are fundamental for the realization of motor body control functions/is not emphasized enough in postural control, within the framework of the ICF activity and participation and the effects on their quality of life has not been sufficiently studied to be a gap in this area, physical/motor control parameters has a significant influence on the body, which is quite activity, participation and quality of life was significantly etkileyecebi it was assumed that their level. In our study, the 6-12 age group was selected because children with Cerebral Palsy at the primary school level have started to become independent from their parents in their daily life activities and have recently adapted to social activities.

In this study, it is aimed to investigate the effect of trunk disorder level on activity, participation and quality of life levels of children with Cerebral Palsy at primary school level.

DETAILED DESCRIPTION:
Cerebral Palsy is a disease characterized by movement, posture and tone disorders that occur in the immature brain structure that has not yet completed its development anatomically and physically, but can undergo permanent changes.Cerebral palsy, neuromuscular diseases and permanent disability among the most widely known throughout the world as the cause of childhood morbidity and mortality rates in takes place at high rates.Many prenatal, perinatal and postnatal problems play a role in the development of Cerebral Palsy. Between Prenatal intrauterine bleeding problems, toxins and infections; perinatal problems between a difficult birth, anoxia; postnatal problems are considered to be among the most frequent causes of premature and low birth weight.

Postural control, which plays a key role in the realization of all our fine and gross motor skills and is necessary for the realization of our daily life activities, is insufficient in children with cerebral palsy, which is a neurological disorder. Insufficient postural control negatively affects mobility, limb movements, static and dynamic trunk control.In recent years, the terms well-being and quality of life have been considered important for the evaluation of health. Well-being is expressed as the well-being of an individual's functional and health condition and an increase in quality of life.SP impaired postural control in children with upper extremity impairment in function, learning difficulties, sensory impairment, dental problems, language-speech disorders, mental retardation, behavior disorders, is illustrated by studies that has a negative impact on quality of life.

When the literature is scanned and trunk postural control more of the physical/motor, we investigated the effect of parameters, which are fundamental for the realization of motor body control functions/is not emphasized enough in postural control, within the framework of the ICF activity and participation and the effects on their quality of life has not been sufficiently studied to be a gap in this area, physical/motor control parameters has a significant influence on the body, which is quite activity, participation and quality of life was significantly etkileyecebi it was assumed that their level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spastic Cerebral Palsy,
* located in the December 7-12 age range,
* Without Severe Mental Retardation,
* GMFCS level 1-2 and 3 are
* Given consent to participate in the study by the parent

Exclusion Criteria:

* Not given consent to participate in the study by the parent,
* Having a type of SP, other than Spastic Cerebral Palsy,
* Severe Mental Retardation and inability to communicate
* not being in the December 7-12 age range -With GMFCS level 4 and 5

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 16 patients with Hemiparetic CP and 16 Diparetic CP will be included.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Trunk Affect Level | First Day
  Static Sitting Balance, Dynamic Sitting Balance and Coordination will be evaluated with the Body Impact Scale (TIS). The scale varies between 0-23 points in total, and high scores indicate that the body control is better.

SECONDARY OUTCOMES:
Activity Level | First Day
  Not to measure the feasibility of the quality of the movement, the international functionality, disability and health as defined in the classification of the 'activity level' and determine tilt, rolling, sitting, crawling, kneeling, standing, walking, jumping, running, containing parameters such as the functional activity of focusing on gross motor function Criteria - GMFM-88 will be assessed.
Level of Participation | First Day
  The functional health status of children and adolescents with CP between the ages of 2-18 will be evaluated by the Pediatric Data Collection Tool (PODCI), which is developed to determine the level of physical function and participation, but also does not ignore the quality of life, answered by parents.
The level of Quality of Life | First Day
  SP-specific developed in order to assess the quality of life, daily activities, school activities, movement and balance, pain and suffering, fatigue, eating, activities, speech and communication, including 7 Sub Module titles for children of cerebral palsy quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Funda ŞEKERCİOĞLU Physiotherapist, Study Chair — Karabuk University; Musa GÜNEŞ MsC, Study Director — Karabuk University; Metehan YANA PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Bourelle S, Berge B, Gautheron V, Cottalorda J. Computerized static posturographic assessment after treatment of equinus deformity in children with cerebral palsy. J Pediatr Orthop B. 2010 May;19(3):211-20. doi: 10.1097/BPB.0b013e32832e957a. PMID 20101192
- [Background] Davis E, Shelly A, Waters E, Davern M. Measuring the quality of life of children with cerebral palsy: comparing the conceptual differences and psychometric properties of three instruments. Dev Med Child Neurol. 2010 Feb;52(2):174-80. doi: 10.1111/j.1469-8749.2009.03382.x. Epub 2009 Jun 22. PMID 19549193
- [Background] Ko J, Kim M. Reliability and responsiveness of the gross motor function measure-88 in children with cerebral palsy. Phys Ther. 2013 Mar;93(3):393-400. doi: 10.2522/ptj.20110374. Epub 2012 Nov 8. PMID 23139425
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Saether R, Helbostad JL, Adde L, Jorgensen L, Vik T. Reliability and validity of the Trunk Impairment Scale in children and adolescents with cerebral palsy. Res Dev Disabil. 2013 Jul;34(7):2075-84. doi: 10.1016/j.ridd.2013.03.029. Epub 2013 May 1. PMID 23643761